CLINICAL TRIAL: NCT05196750
Title: Effect of Obstetric Anesthesia and Delivery Mode On Neurodevelopmental And Behavioural Outcomes In A Population-Based Birth Cohort
Status: Completed | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: CIRB 2021/2113
Record Dates: First submitted 2021-10-24; First posted 2022-01-19 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-06

CONDITIONS: Neurodevelopmental Disorders; Behavior
Keywords: Obstetric Anaesthesia
MeSH Terms: conditions — Neurodevelopmental Disorders; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal vaginal delivery: Maternal delivery of delivery via normal vaginal delivery
  Interventions: Other: Behavioural questionnaires and assessments on mother and child
- Lower segment Caesarean section (LSCS): Maternal delivery of delivery via lower segment Caesarean section (LSCS)
  Interventions: Other: Behavioural questionnaires and assessments on mother and child

INTERVENTIONS:
Other: Behavioural questionnaires and assessments on mother and child — Questionnaires include, but not limited to, State Trait Anxiety Inventory, Beck Depression Inventory, LYNDON Maternal Health and Well Being, Facial Imitation Task, Deferred Imitation, Habituation, Relational Binding, Behavioural Observation, Mirror Self Recognition, Standardized Assessment and Experimental Task, Snack and Sticker Delay, Implicit Attitude Test

SUMMARY:
The study aims to determine:

1. The association between Obstetric anesthesia events at delivery (such as mode of anesthesia, drugs given, desaturation and hypotension) on pediatric neurodevelopmental and behavioural outcomes.
2. Mode of delivery on pediatric neurodevelopmental and behavioural outcomes.
3. Effect of labour epidural analgesia on neurodevelopmental and behavioural outcomes.
4. To determine if these would differ between very preterm, moderate preterm, late preterm and term infants.

The study team hypothesise that:

1. Adverse maternal events during anesthesia and labor analgesia may be associated with poorer neurodevelopmental outcomes in infants.
2. Delivery via a lower segment caesarean section (LSCS) combined with a general anesthetic during delivery may be associated with adverse pediatric neurodevelopmental and behavioural outcomes.
3. The use of labour epidural analgesia is associated with poorer neurodevelopmental and behavioural outcomes.
4. These differences may be more pronounced in preterm infants as compared to term infants.

DETAILED DESCRIPTION:
The relationship between the mode of delivery, type of anesthesia received, maternal anesthetic events at delivery and its effects on pediatric neurodevelopment and behavioral outcomes remains poorly defined with previous work showing conflicting results. Furthermore, previous studies have failed to take into account the potential effect of other antepartum anesthetic events such as the type of anesthesia, hypotension or desaturation. Furthermore, majority have failed to stratify between the subsets of premature infants, who may inherently be more susceptible to neurodevelopmental insult.

The GUSTO study is well-placed to provide unique insight with regards to these domains, due to its comprehensive, sensitive and specific follow-up of pediatric neurocognitive development and in-depth maternal anesthetic delivery data. Hence, previously collected, existing data from the Growing Up in Singapore Towards healthy Outcomes (GUSTO) cohort study will be utilized for this study.

This will be supplemented by additional maternal anesthetic and delivery data which the investigators aim to collect via a retrospective chart review.

ELIGIBILITY:
Inclusion Criteria:

* All mothers and infants recruited into the GUSTO database from 2011 to 2016, who underwent neurodevelopmental follow-up will be included in the study.

Exclusion Criteria:

* Children who dropped out of the study before 18 months of age
* Children who had subsequent exposure to general anaesthesia/surgeries/sedatives

Ages: 0 Years to 10 Years | Sex: All
Age Groups: Child
Study Population: All mothers and infants recruited into the GUSTO database from 2011 to 2016, who underwent neurodevelopmental follow-ups.
Sampling Method: Non-Probability Sample
Enrollment: 1176 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
Association between Obstetric anesthesia events at delivery on pediatric neurodevelopmental and behavioural outcomes via questionnaires administered | Prenatal to postnatal up to 7 years
  To establish an association with the prenatal, antenatal and postnatal data previously collected in the GUSTO study.
Mode of delivery on pediatric neurodevelopmental and behavioural outcomes via questionnaires administered | Prenatal to postnatal up to 7 years
  Trend neurodevelopmental outcomes between infants born from normal vaginal delivery and LSCS.
Effect of labour epidural analgesia on neurodevelopmental and behavioural outcomes via questionnaires administered | Prenatal to postnatal up to 7 years
  Trend neurodevelopmental outcomes between infants born from normal vaginal delivery and LSCS.

CONTACTS AND LOCATIONS:
Overall Officials: Choon Looi Bong, Principal Investigator — KKH Women and Children's Hospital
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore
  - KKH Women and Children Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sprung J, Flick RP, Wilder RT, Katusic SK, Pike TL, Dingli M, Gleich SJ, Schroeder DR, Barbaresi WJ, Hanson AC, Warner DO. Anesthesia for cesarean delivery and learning disabilities in a population-based birth cohort. Anesthesiology. 2009 Aug;111(2):302-10. doi: 10.1097/ALN.0b013e3181adf481. PMID 19602960
- [Background] Chen G, Chiang WL, Shu BC, Guo YL, Chiou ST, Chiang TL. Associations of caesarean delivery and the occurrence of neurodevelopmental disorders, asthma or obesity in childhood based on Taiwan birth cohort study. BMJ Open. 2017 Sep 27;7(9):e017086. doi: 10.1136/bmjopen-2017-017086. PMID 28963295
- [Background] Curran EA, O'Neill SM, Cryan JF, Kenny LC, Dinan TG, Khashan AS, Kearney PM. Research review: Birth by caesarean section and development of autism spectrum disorder and attention-deficit/hyperactivity disorder: a systematic review and meta-analysis. J Child Psychol Psychiatry. 2015 May;56(5):500-8. doi: 10.1111/jcpp.12351. Epub 2014 Oct 27. PMID 25348074
- [Background] Qiu C, Lin JC, Shi JM, Chow T, Desai VN, Nguyen VT, Riewerts RJ, Feldman RK, Segal S, Xiang AH. Association Between Epidural Analgesia During Labor and Risk of Autism Spectrum Disorders in Offspring. JAMA Pediatr. 2020 Dec 1;174(12):1168-1175. doi: 10.1001/jamapediatrics.2020.3231. PMID 33044486